CLINICAL TRIAL: NCT04375982
Title: A Multicenter Study Conducted to Evaluate the Agreement Between Fingerstick Whole Blood, Venous Whole Blood and Plasma Determined on the LumiraDx Point of Care D-Dimer and Point of Care CRP Tests to Results on the Reference Analyzer
Brief Title: Evaluation of the LumiraDx Point of Care D-Dimer and CRP Tests
Acronym: NOVEL-3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-CLIN-PROT-00027
Record Dates: First submitted 2020-04-30; First posted 2020-05-06 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Embolism and Thrombosis; Infection; Inflammation
MeSH Terms: conditions — Embolism and Thrombosis; Infections; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Subjects are asked to provide venous and capillary blood samples which are not being taken as part of routine care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Blood collection (Other): Venepuncture and fingerstick to obtain venous blood and capillary blood respectively
  Interventions: Diagnostic Test: Venepuncture; Diagnostic Test: Fingerstick

INTERVENTIONS:
Diagnostic Test: Venepuncture — Blood tube will be collected from standard venepuncture
Diagnostic Test: Fingerstick — Capillary blood will be collected by fingerstick

SUMMARY:
A Multicenter Study Conducted to Evaluate the Agreement between Fingerstick Whole Blood, Venous Whole Blood and Plasma Determined on the LumiraDx Point of Care D-Dimer and Point of Care CRP Tests to Results on the Reference Analyzer

DETAILED DESCRIPTION:
The purpose of the study is to gather data to determine agreement between sample types, which together with performance evaluation data will be used to support CE marking under Directive 98/79/EC of the European Parliament and of the Council of 27 October 1998 on in vitro diagnostic medical devices 3, using ISO 13612:2002 - Performance Evaluation of In Vitro Diagnostic Medical Devices as the standard. The investigative devices are the LumiraDx Platform D Dimer Test and the LumiraDx Platform CRP Test. The LumiraDx Platform employs a portable diagnostic instrument used with single use D Dimer or CRP Assay Test Strips.

Agreement of the different sample types to the reference method will be demonstrated across a patient population representative of the indication for use of the products. Operators will be trained clinical site staff who are representative of the intended users of the product, i.e. health care professionals at the point of care such as nurses, technicians, doctors, etc. A panel of whole blood and plasma samples will be obtained from each patient in order to assess the accuracy of the investigative device across all sample types.

ELIGIBILITY:
Inclusion Criteria D-dimer:

* Subjects >18 years of age.
* Willing and able to provide written informed consent and comply with study procedures.
* Presenting to healthcare provider for any reason* *All presentations are suitable for recruitment; however, the following conditions are of particular interest: Venous thromboembolism symptoms (DVT and Pulmonary embolism), subjects seeking medical attention with symptoms of respiratory tract infection (upper or lower), Acute myocardial infarction / unstable angina, Anti-inflammatory medication (current), Any regular medication for a chronic condition (other than simple painkiller or inhaler), Atrial fibrillation, Diabetes mellitus (all types except 'pre-diabetes'), Heart failure, Hypertension (>150/90), Infection (significant current or within 3 months), Peripheral arterial disease, Surgery (within 6 weeks), Childbirth (within 8 weeks), Significant trauma, burns (within 4 weeks), Pregnancy (confirmed or suspected), Acute upper gastrointestinal haemorrhage other significant recent haemorrhage.

D-dimer Exclusion Criteria:

* The subject is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic or drug including either treatment or therapy.
* Skin lesions or conditions that would preclude a fingerstick and or a venous blood draw.
* End-stage renal failure on haemodialysis.
* Life expectancy documented as less than 30 days.
* Haemodynamically unstable (e.g. cardiogenic shock).
* Current anticoagulation therapy (Fragmin, LMWH) within the last 30 days.
* Patients taking anticoagulant therapy (DOACS, Warfarin, Heparins etc.) within the last 30 days.
* The subject has previously participated in this research study

CRP Inclusion criteria:

* Subjects >18 years of age.
* Willing and able to provide written informed consent and comply with study procedures.
* Subjects seeking medical attention with symptoms of infection, tissue injury, inflammatory disorders or associated disease. This includes but not limited to: respiratory tract infection (upper or lower), rheumatoid arthritis, Lupus, burns, trauma, inflammatory bowel disease.

CRP Exclusion Criteria:

* The subject is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic or drug including either treatment or therapy.
* Skin lesions or conditions that would preclude a fingerstick and or a venous blood draw.
* A subject with a critical illness, requiring critical intervention, or end of life or palliative care.
* Subjects suffering with Myeloma, Monoclonal Gammopathy or extreme Lipaemia.
* The subject has previously participated in this research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of sample matrix comparison | 2 months
  Verification that all sample types give an equivalent result when tested in the LumiraDx assays. Results generated from capillary blood and venous whole blood will be compared to those generated from plasma to ensure that all 3 sample types give equivalent values. Results will be compared by standard statisitical techniques which may include Regression analysis (e.g. Passing Bablok) or Bias analysis (e.g. Altman Bland)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Kirstein, Principal Investigator — Rancho Paseo Medical Group; Matthew Morgan, Principal Investigator — Centura Health Physician Group; Anita Scribner, Principal Investigator — Diagnostic Clinic of Longview; William Simon, Principal Investigator — New Medical Healthcare
Locations (4):
- United States (4):
  - Rancho Paseo Medical Group, Banning, California
  - Centura Health Physician Group, Northglenn, Colorado
  - New Medical Healthcare, Wichita, Kansas
  - Diagnostic Clinic of Longview, Longview, Texas

IPD SHARING:
Plan to Share IPD: No